CLINICAL TRIAL: NCT06589973
Title: IImpact of Clinical and Biochemical Variables on Mortality and Morbidity of Patients With Alcohol Withdrawal Syndrome Under Treatment According to the CIWA-AR Scale"
Brief Title: Effect of Clinical and Biochemical Variables Over Morbidity and Mortality in Alcohol Withdrawal Syndrome Patients
Status: Recruiting | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Principal investigator, Hospital General de Mexico
Other Study IDs: 606023-01-1624
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Withdrawal Syndrome
MeSH Terms: interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study Cohort — Clinical records (files) of patients with a diagnosis of admission of alcohol withdrawal syndrome (AAS) who have been treated in the Department of Internal Medicine for 5 years.

SUMMARY:
The goal of this observational study is to describe the impact measured through the Odds Ratio (OR) of different variables of clinical and biochemical alterations on the duration of the syndrome alcohol withdrawal patients measured in days of symptoms and stay; it could include any patients with a diagnosis of admission of alcohol withdrawal syndrome (AWS) who have been treated in the department of Internal Medicine for 5 years.

The main question it aims to answer is: What is the relationship between the different clinical, biochemical, and hematic factors on the duration of symptoms, morbidity, and mortality in individuals with alcohol syndrome withdrawal?

• If the patient has a greater number of risk factors, such as advanced age, a long and chronic history of alcohol consumption, the type of distillate consumed, as well as the deterioration of liver function and presence of leukocytosis and neutrophilia, then it is postulated that the duration of alcohol withdrawal syndrome will be longer.

Clinical records will be used to describe the proportion of complications associated with alcohol withdrawal syndrome including pneumonia bronchial aspiration, seizures, need for mechanical ventilation, digestive tract hemorrhage, toxic-alcoholic hepatitis, and pancreatitis.

DETAILED DESCRIPTION:
Clinical records (files) of patients with a diagnosis of admission of alcohol withdrawal syndrome (AAS) who have been treated in the Department of Internal Medicine for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical records of patients, both genders, over 18 years of age with Alcohol Withdrawal Syndrome according to the criteria for alcohol withdrawal.
* Clinical records of candidates for admission for neurological monitoring and with criteria for use of sedative drugs according to the CIWA-Ar scale
* Clinical records of patients containing the CIWA-Ar scale score at diagnosis

Exclusion Criteria:

* Clinical records of patients who already have a history of seizures or epilepsy
* Clinical records of diabetic patients with diabetic ketoacidosis
* Clinical records of patients who have not received any type of sedative treatment
* Clinical records of patients with chronic liver failure or liver cirrhosis
* Clinical records of patients with chronic liver disease with signs of hepatic encephalopathy
* Clinical records of patients with related toxic-alcoholic hepatitis
* Clinical records of patients with a life expectancy of less than 24 hours due to associated complications such as head trauma or other associated complications
* Clinical records of patients who require intubation and mechanical ventilation upon admission
* Clinical records of patients who have a vascular event that modifies the neurological evaluation
* Clinical records of patients who before admission show psychomotor alteration or neurological deterioration that modifies the neurological evaluation such as the presence of Wernicke's encephalopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical records (case files) of patients with an admission diagnosis of alcohol withdrawal syndrome (AWS) who have been treated in the Internal Medicine department for 5 years will be analyzed.
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Death | 6 months
  Permanent cessation of all vital functions of an organism, including irreversible stopping of the heart and breathing
Morbidity | 6 months
  Any type of complication present during the analysis period that complicates the resolution of the condition, including serious situations.

SECONDARY OUTCOMES:
Hospital stay | 6 months
  Time recorded in the clinical record of the duration of symptoms from the first clinical manifestation until the time of discharge.
Duration of symptoms | 6 months
  Time recorded in the clinical record of the duration of symptoms from the first clinical manifestation to the description of improvement in the medical notes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Cuautitlan "General José Vicente Villada", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Due to privacy and confidentiality restrictions, the data presented in this study is available on request from the corresponding author. The data are not publicly available due to the confidentiality restrictions of the Biosecurity, Ethics, and Research Committee of Hospital General de Cuatitlan "General José Vicente Villada"